CLINICAL TRIAL: NCT04538794
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Multiple Ascending Dose Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of CDX-0159 as Add-on Therapy in Patients With Chronic Spontaneous Urticaria
Brief Title: A Study of CDX-0159 in Patients With Chronic Spontaneous Urticaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDX0159-02; 2020-005426-29 (EudraCT Number)
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: CDX-0159
MeSH Terms: conditions — Chronic Urticaria | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CDX-0159 (Experimental): CDX-0159 every 4-8 weeks
  Interventions: Drug: CDX-0159
- Normal Saline (Placebo Comparator): Normal saline every 4-8 weeks
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: CDX-0159 — Administered intravenously
  Arms: CDX-0159
Drug: Normal Saline — Administered intravenously
  Arms: Normal Saline

SUMMARY:
This is a study to determine the safety of multiple doses of CDX-0159 in patients with Chronic Spontaneous Urticaria.

DETAILED DESCRIPTION:
The purpose of the study is to explore the safety, pharmacodynamics, and pharmacokinetics of ascending doses of CDX-0159 in patients with Chronic Spontaneous Urticaria who remain symptomatic despite treatment with antihistamines.

There is a screening period of up to 2 weeks, a 12-week double-blind treatment period and a 12-week follow-up period after treatment. Patients will receive multiple doses of CDX-0159 or placebo as add on therapy to their antihistamine.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females, 18 - 75 years old.
2. Diagnosis of chronic spontaneous urticaria (CSU) despite the use of H1-antihistamines alone or in combination with H2-antihistamines and/or leukotriene receptor antagonists, as defined by:

   1. Diagnosis of CSU for >/= 6 months.
   2. The presence of itch and hives for >/= 6 consecutive weeks at any time prior to Visit 1 despite current use of H1-antihistamines.
   3. UAS7 of >/= 16 and HSS7 of >/= 8 during the 7 days before treatment
   4. In-clinic UAS >/= 4 on one of the screening visit days
   5. Use of H1-antihistamines alone or in combination with H2-antihistamines and/or leukotriene receptor antagonists for at least 3 days immediately prior to study entry and throughout the study.
3. Other than CSU, have no other significant medical conditions that would cause additional risk or interfere with study procedures.
4. Normal blood counts and liver function tests.
5. Both males and females of child-bearing potential must agree to use highly effective contraceptives during the study and for 150 days afterwards after treatment.
6. Willing and able to complete a daily symptom electronic diary for the duration of the study and adhere to the study visit schedule.

Key Exclusion Criteria:

1. Women who are pregnant or nursing.
2. Cleary defined cause for chronic urticaria.
3. Known HIV, hepatitis B or hepatitis C infection.
4. Vaccination with a live vaccine within 4 weeks prior to study drug administration (subjects must agree to avoid vaccination during the study). Inactivated vaccines are allowed such as seasonal influenza for injection.
5. History of anaphylaxis.

There are additional criteria that your study doctor will review with you to confirm you are eligible for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by the incidence and severity of adverse events | From Day 1 (first dose) to Day 169 (last follow-up visit)
  Safety of multiple, ascending doses of CDX-0159 as determined by drug related adverse events

SECONDARY OUTCOMES:
Pharmacokinetic evaluation | From Day 1 (before first dose) to Day 169 (last follow-up visit)
  CDX-0159 serum concentrations will be measured at specified visits
Pharmacodynamic evaluation | From Day 1 (first dose) to Day 169 (last follow-up visit)
  The change from baseline for Urticaria Activity Score (UAS7) in patients who received CDX-0159 vs. placebo
Pharmacodynamic evaluation | From Day 1 (first dose) to Day 169 (last follow-up visit)
  The change from baseline for Hives Severity Score (HSS7) in patients who received CDX-0159 vs. placebo
Pharmacodynamic evaluation | From Day 1 (first dose) to Day 169 (last follow-up visit)
  The change from baseline for Itch Severity Score (ISS7) in patients who received CDX-0159 vs. placebo
Pharmacodynamic evaluation | Day 1 (first dose) to Day 169 (last follow up visit)
  The change in baseline for Urticaria Control Test (UCT) in patients who received CDX-0159 vs. placebo
Pharmacodynamic evaluation | From Day 1 (before first dose) to Day 169 (last follow-up visit)
  The effect of CDX-0159 on stem cell factor levels
Pharmacodynamic evaluation | From Day 1 (before first dose) to Day 169 (last follow-up visit)
  The effect of CDX-0159 on tryptase
Safety evaluation | From Day 1 (before dosing) to Day 169 (last follow-up visit)
  Assessment of immunogenicity by measuring the development of anti- CDX-0159 antibodies

CONTACTS AND LOCATIONS:
Locations (14):
- United States (13):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Arizona Allergy & Immunology Research, Gilbert, Arizona
  - Sarasota Clinical Research, Sarasota, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Midwest Allergy, Sinus and Asthma, SC, Normal, Illinois
  - Dawes Fretzin Clinical Research, Indianapolis, Indiana
  - Kanarek Allergy Asthma & Immunology, Overland Park, Kansas
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Asthma, Nasal Disease & Allergy Research Center of New England, East Providence, Rhode Island
  - National Allergy and Asthma Research, LLC, North Charleston, South Carolina
  - AARA Research, Dallas, Texas
- Charite University, Berlin, Germany